CLINICAL TRIAL: NCT04207138
Title: To Study the Association Among Labor Pain and Physical Parameters in Laboring Pregnant Women
Status: Withdrawn | Type: Observational
Why Stopped: change sponsor
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201910058RIPC
Record Dates: First submitted 2019-12-17; First posted 2019-12-20 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2019-12

CONDITIONS: Labor Pain
Keywords: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Analysis of monitored clinically parameters during the course of labor is a seldom studied area in Taiwan and worldwide. Important monitored parameters include, fetal heartbeat, uterine contractions, oxygen saturation and blood pressure, among others.1 During labor, uterine contractions can cause pain.3 This pain may be measured using a visual analogue scale (VAS).2 The pain from uterine contractions promotes the release of hormones including cortisol which can cause decreased or irregular contractions and possibly prolong labor.3 This study aims to study the association between monitored clinical parameters and pain in women in Taiwan during labor in order to increase the understanding to safe childbirth.

DETAILED DESCRIPTION:
This is a prospective, observational study to measure and collect and physical parameters from females at least 20 years of age in the labor room. Collection of measurements and physical parameters will begin when the subject enrolls in the study. Besides, ECG and SpO2 will be recorded continuously until the end of the study period. In addition, uterus contraction cycle and fetal heart beat will be recorded during the study period based on standard of care in the labor room. Pain will be recorded on a visual analogue scale (VAS) at baseline and when the caregiver perceives that there is a change in the subject's pain status until the end of the study period. The time of each assessment of pain on VAS should be recorded. Subjects will be withdrawn from the study if they have a cesarean section or any complication during labor in the opinion of the investigator. Subject participation in the study will end when eight hours have elapsed since baseline, the subject leaves the labor room or the subject delivers the baby.

ELIGIBILITY:
Inclusion criteria:

1. Female at least 20 years of age.
2. Have a course of labor that is > 4 hours.
3. American Society of Anesthesiologists Physical Status (ASA PS) Classification of Class I-II.
4. Clinical records of the subject are complete in the opinion of the investigator.

Exclusion criteria:

1. Subject has any condition, which in the opinion of the investigator precludes the subject's participation in the study.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Maternity at least 20 years of age in the labor room
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-04-14 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
To detect the association between labor pain and related physical parameters during labor progression | Eight hours have elapsed since baseline or the subject leaves the labor room or the subject delivers the baby
  Collection of measurements and physical parameters will begin when the subject enrolls in the study. Besides, ECG and SpO2 will be recorded continuously until the end of the study period. In addition, uterus contraction cycle and fetal heart beat will be recorded during the study period based on standard of care in the labor room. Pain will be recorded on a visual analogue scale (VAS) at baseline and when the caregiver perceives that there is a change in the subject's pain status until the end of the study period. The time of each assessment of pain on VAS should be recorded. Subjects will be withdrawn from the study if they have a cesarean section or any complication during labor in the opinion of the investigator. Subject participation in the study will end when eight hours have elapsed since baseline, the subject leaves the labor room or the subject delivers the baby.

CONTACTS AND LOCATIONS:
Overall Officials: CHIEN-NAN LEE, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan